CLINICAL TRIAL: NCT01597557
Title: Intravenous Magnesium Infusion in Patients Undergoing Cardioversion of Atrial Fibrillation Trial
Acronym: MICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Anne Curtis, Principal investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MED7441011B
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Electrical Cardioversion; Magnesium Sulfate
MeSH Terms: conditions — Atrial Fibrillation | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium Sulfate (Active Comparator): Patients in this arm are give magnesium sulfate 2 grams intravenous drip before the cardioversion procedure
  Interventions: Drug: Magnesium Sulfate
- Placebo (Placebo Comparator): Patients in this arm receive normal saline drip intravenously before the cardioversion procedure
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Magnesium Sulfate — 2 grams intravenous drip over 30 minutes
  Arms: Magnesium Sulfate
Other: Placebo — Normal Saline 50 ml intravenous drip over 30 minutes
  Arms: Placebo

SUMMARY:
The proposed study is designed to evaluate the effect of an intravenous infusion of magnesium sulfate in facilitating successful cardioversion of atrial fibrillation and in decreasing the energy threshold (in J) required for successful cardioversion of atrial fibrillation into sinus rhythm.

DETAILED DESCRIPTION:
Patients with atrial fibrillation may suffer from disabling symptoms such as palpitations, shortness of breath or worsening heart failure. In such patients, it may be beneficial to convert their rhythm to sinus rhythm. Cardioversion can be achieved either pharmacologically or electrically. Pharmacological cardioversion is less successful acutely than electrical cardioversion and may be associated with complications such as prolongation of the QT interval and torsades de pointes (polymorphic ventricular tachycardia). Thus, cardioversion is most often accomplished electrically, using biphasic synchronized shocks of 75-200 Joules. Biphasic electrical cardioversion in atrial fibrillation has shown to be successful (i.e., converting to sinus rhythm) about 88% of the time, on average. The success rate appears to largely depend upon the duration of the arrhythmia and the presence and severity of structural heart disease.

In this study, we will evaluate the effect of intravenous magnesium sulfate on the success rate of electrical cardioversion, and also assess its effect in decreasing the energy levels needed for successful cardioversion. If the study is successful, we will have shown that a simple and inexpensive intervention can increase the success rate of electrical cardioversion, increasing the proportion of patients who can be restored to sinus rhythm. In addition, success with lower energy levels may improve the safety of cardioversion, as high energy levels are more likely to be associated with side effects

ELIGIBILITY:
Inclusion Criteria:

* Patient with new onset Atrial fibrillation less than 48 hours after onset undergoing electrical cardioversion.
* Patients with atrial fibrillation longer than 48 hours on warfarin with documented therapeutic INR levels >2 for at least 3 weeks prior to the cardioversion, or been on dabigatran for 3 weeks, or a transesophageal echocardiogram on the day of the procedure that excludes intracardiac thrombi, undergoing electrical cardioversion.

Exclusion Criteria:

* Creatinine >2.0 mg/dl
* Potassium level less than 3.5 mmol/dl
* TSH < 0.5
* Magnesium levels >3.0 mg/dl
* Urgent need for cardioversion (e.g., hemodynamic instability, unstable angina, pulmonary edema)
* Patients with recent (less than 6 weeks) acute myocardial infarction
* Patients post-cardiac surgery
* Pregnant women
* Patients who are being treated with antiarrhythmic drugs who have received less than five doses of the drug. For amiodarone, patients who have received less than three weeks prior to cardioversion are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2012-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne B Curtis, MD, Principal Investigator — State University of New York at Buffalo; Bharath Rajagopalan, MBBS, Principal Investigator — State University of New York at Buffalo; Anne B Curtis, MD, Study Chair — State University of New York at Buffalo
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Derived] Rajagopalan B, Shah Z, Narasimha D, Bhatia A, Kim CH, Switzer DF, Gudleski GH, Curtis AB. Efficacy of Intravenous Magnesium in Facilitating Cardioversion of Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2016 Sep;9(9):e003968. doi: 10.1161/CIRCEP.116.003968. PMID 27586232

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some patients enrolled in the study and received the study drug but did not undergo the cardioversion procedure due to various reasons
Period: Overall Study
Arm/Group | Magnesium Sulfate | Placebo
Started | 132 | 129
Completed | 128 | 126
Not Completed | 4 | 3
Not completed — Did not undergo cardioversion procedure | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Sulfate | Placebo | Total
Number analyzed (Participants) | 132 | 129 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.4) | 65.6 (11.9) | 65.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 38 | 81
  Male | 89 | 91 | 180
Region of Enrollment [Number; unit: participants]
  United States | 132 | 129 | 261

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Cardioversion of Atrial Fibrillation to Sinus Rhythm
Description: Successful cardioversion involves conversion of atrial fibrillation to sinus rhythm and maintenance of sinus rhythm for one hour
Time Frame: One hour after cardioversion
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium Sulfate | Placebo
Number analyzed (Participants) | 132 | 129
Participants | 114 | 111

2. Secondary Outcome: Total Amount of Energy Required for Successful Cardioversion of the Atrial Fibrillation to Sinus Rhythm
Time Frame: One hour
Population: Some patients enrolled in the study and received the study drug but did not undergo the cardioversion procedure per protocol and were excluded in this analysis
Measure: Mean (Standard Deviation); unit: Joules
Arm/Group | Magnesium Sulfate | Placebo
Number analyzed (Participants) | 130 | 126
Joules | 123.3 (55.5) | 129.5 (52.6)

3. Secondary Outcome: Number of Participants Who Experienced Severe Hypotensive Episodes After Infusion of Magnesium Sulfate or Placebo
Description: Severe hypotensive episode with a Systolic BP < 90mm hg with > 20 mm Hg drop after infusion of the study drug or placebo
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium Sulfate | Placebo
Number analyzed (Participants) | 132 | 129
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Magnesium Sulfate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/129
Other Adverse Events (participants affected / at risk) | 0/132 | 0/129

LIMITATIONS AND CAVEATS:
Very few patients in paroxysmal AF, majority failed earlier rhythm control strategies making the study population a resistant population to treat, only one dose of Mg infusion was tested and the monitoring period was only 1 hour post cardioversion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No